CLINICAL TRIAL: NCT04421742
Title: The Effect of Beclomethasone/Formoterol in Extra-fine Formulation on Quality of Life and Dyspnea is Associated to the Improvement in Small Airway Dysfunction in COPD Patients. A Pilot Study (IOSCOPD20161102)
Brief Title: The Effect of Beclomethasone/Formoterol in Extra-fine Formulation on Quality of Life and SAD in COPD Patients.
Status: Completed | Type: Observational
Sponsor: Alfredo Antonio Chetta (Other)
Collaborators: University of Parma (Other)
Responsible Party: Sponsor-Investigator, Alfredo Antonio Chetta, Clinical Professor, University of Parma
Organization: University of Parma (Other)
Other Study IDs: 9769 del 15.03.2017
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 43 COPD: COPD patients with severe airflow obstruction and 1 moderate exacerbation in the previous year being treated with BDP/FF NEXThaler® 100/6 μg b.i.d. for 12 weeks
  Interventions: Drug: Beclomethasone Dipropionate/Formoterol Fumarate

INTERVENTIONS:
Drug: Beclomethasone Dipropionate/Formoterol Fumarate — BDP/FF NEXThaler® 100/6 μg b.i.d.
  Other Names: Foster NEXThaler®

SUMMARY:
In patients with chronic obstructive pulmonary disease (COPD), small-airway dysfunction (SAD) is considered a key element and a functional consequence of the pathology. However, the exact role of SAD as a specific 'pharmacological target' is not yet fully known.

Objectives In an open-label prospective study, we aimed to ascertain whether an extra-fine formulation of Beclomethasone dipropionate/Formoterol fumarate (BDP/FF) NEXThaler® 100/6 μg b.i.d. can improve the impact of the disease on the quality of daily life of COPD patients, acting on SAD.

Methods We studied COPD patients with severe airflow obstruction and 1 moderate exacerbation in the previous year, being treated with BDP/FF NEXThaler® for 12 weeks. They underwent three visits, at the start of the treatment (V1), at 6th week (V2) and at 12th week (V3). By the impulse oscillometry system and by spirometry and plethysmography we measured at each visit the fall in resistance from 5 to 20 Hz (R5-R20) and the residual volume/total lung capacity (RV/TLC). COPD Assessment Test (CAT) and the modified Medical Research Council (mMRC) questionnaire were also measured at each visit to assess the impact of the disease on the quality of life of the patients.

DETAILED DESCRIPTION:
In recent years, there has been a growing interest in deepening the contribution of small airways (with a diameter <2mm) to the clinical expression of Chronic Obstructive Pulmonary Disease (COPD).

In patients with stable COPD, SAD severity was found to be progressively increased both with the degree of airflow obstruction and with GOLD risk class. Moreover, a correlation between SAD and COPD impact measured with the CAT (COPD Assessment Test) was found, being the severity of SAD a predictor of the impact of the disease (CAT≥10). A close correlation between SAD and both quality of life (measured with the St. George's Respiratory Questionnaire) and perceived dyspnea (measured with the modified Medical Research Council-mMRC scale) was also found in COPD patients.

The exact role of SAD as a specific 'pharmacological target' is not yet fully known. According to the guidelines, the administration of combination such as Beclomethasone dipropionate/Formoterol fumarate (BDP/FF) in extra-fine formulation produced a clinically relevant improvement in quality of life (> 4 units in the St. George's Respiratory Questionnaire) and in dyspnea. However, it is not yet defined whether exists a correlation between symptomatic improvement and SAD and whether an improvement of symptoms can be achieved acting pharmacologically on SAD.

The rationale for this study is based on the hypothesis that an extra-fine formulation of BDP/FF, designed to target the entire bronchial three, included the peripheral zone, can improve the impact of the disease on the quality of life of COPD patients, acting on SAD. The functional indices of SAD used in this study are from the impulse oscillometry system (IOS), the standard spirometry and the body plethysmography.

The primary endpoint of the study was, therefore, an improvement of the impact of the disease on quality of daily life (CAT) and of dyspnea (mMRC) after 12th week treatment with an extra-fine formulation of BDP/FF in a cohort of COPD patients with severe airway obstruction and one moderate exacerbation in a previous year; secondary endpoint was an improvement of the SAD at the 12th week in these patients.

ELIGIBILITY:
Inclusion Criteria:

* a documented diagnosis of COPD defined according to the guidelines of the American Thoracic Society (ATS) / European Respiratory Society (ERS);
* smokers or former smokers with a smoking history of at least 10 pack / years;
* subjects with a post-bronchodilator forced expiratory volume at the 1st second (FEV1)/ forced vital capacity (FVC) ratio of < 0.7 and a FEV1 <50% pred;
* subjects with a high impact of the COPD on their health status (CAT≥10);
* clinical history of at least 1 moderate exacerbation / year;
* COPD patients being treated with BDP/FF NEXThaler® 100/6 μg in extra-fine formulation no more than 1 (one) week before enrollment.

Exclusion Criteria:

* an exacerbation in the four weeks prior to enrollment;
* other coexisting lung diseases (bronchial asthma, restrictive diseases or bronchiectasis) and severe co-morbidities associated with COPD, such as uncontrolled cardiovascular disease, pneumonia or cancer;
* pregnant patients;
* subjects unable to meet the criteria of acceptability and repeatability of pulmonary function tests, according to the ATS / ERS document

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients of the outpatient clinic of the Respiratory Disease Unit of the University Hospital in Parma (Italy)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Change (Improvement) of CAT (Italian version) | Change from Baseline CAT at 12th week
  The CAT (COPD Assessment Test) is a questionnaire suitable for completion by all patients diagnosed with COPD. It comprises 8 simple questions that most patients should be able to understand and complete independently.
  The CAT has a scoring range of 0-40, where each question is ranging 0-5. A CAT score>10 indicates a medium/high impact level of COPD.
  A difference or change of 2 or more units over 2 to 3 months in a patient suggests a clinically significant difference or change in health status (minimal clinically relevant change, often referred to as the Minimum Clinically Important Difference or MCID).
Change (Improvement) of mMRC (Italian version) | Change from Baseline mMRC at 12th week
  The modified Medical Research Council (mMRC) dyspnoea scale is a questionnaire that consists of five statements about perceived breathlessness: grade 1, "I only get breathless with strenuous exercise"; grade 2, "I get short of breath when hurrying on the level or up a slight hill"; grade 3, "I walk slower than people of the same age on the level because of breathlessness or have to stop for breath when walking at my own pace on the level"; grade 4, "I stop for breath after walking 100 yards or after a few minutes on the level"; grade 5, " I am too breathless to leave the house". Patients are asked about their perceived breathlessness and are then classified into MRC dyspnoea grades according to how they perceive their disability.
Change (Improvement) of R5-R20 (kPa x s x L-1) | Change from Baseline R5-R20 at 12th week
  The IOS was performed with the Jaeger MasterScreen-IOS device following the standard recommendations. Respiratory resistances at 5 Hz and 20 Hz (R5 and R20, kPa x s x L-1) were used as a total and proximal airway resistance index, respectively, and the resistance drop from 5 to 20 Hz (R5 - R20, kPa x s x L-1) was considered as an indirect index of resistance of the peripheral airways. The oscillometer was calibrated daily.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo A Chetta, MD, Principal Investigator — Hospital-University of Parma, Italy
Locations (1):
- Department of Medicine and Surgery, Respiratory Disease and Lung Function Unit, University of Parma, Italy, Parma, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected in this study are available to other researches
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available starting from 6 months after publication
Access Criteria: Data will be shared with the Principal Investigator and the authors, if requested, by e-mail contacting
URL: http://unipr.it

REFERENCES:
- [Result] Burgel PR. The role of small airways in obstructive airway diseases. Eur Respir Rev. 2011 Mar;20(119):23-33. doi: 10.1183/09059180.00010410. PMID 21357889
- [Result] Hogg JC, Chu F, Utokaparch S, Woods R, Elliott WM, Buzatu L, Cherniack RM, Rogers RM, Sciurba FC, Coxson HO, Pare PD. The nature of small-airway obstruction in chronic obstructive pulmonary disease. N Engl J Med. 2004 Jun 24;350(26):2645-53. doi: 10.1056/NEJMoa032158. PMID 15215480
- [Result] Crisafulli E, Pisi R, Aiello M, Vigna M, Tzani P, Torres A, Bertorelli G, Chetta A. Prevalence of Small-Airway Dysfunction among COPD Patients with Different GOLD Stages and Its Role in the Impact of Disease. Respiration. 2017;93(1):32-41. doi: 10.1159/000452479. Epub 2016 Nov 17. PMID 27852080
- [Result] Wedzicha JA, Singh D, Vestbo J, Paggiaro PL, Jones PW, Bonnet-Gonod F, Cohuet G, Corradi M, Vezzoli S, Petruzzelli S, Agusti A; FORWARD Investigators. Extrafine beclomethasone/formoterol in severe COPD patients with history of exacerbations. Respir Med. 2014 Aug;108(8):1153-62. doi: 10.1016/j.rmed.2014.05.013. Epub 2014 Jun 6. PMID 24953015
- [Result] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Result] George J, Kong DC, Thoman R, Stewart K. Factors associated with medication nonadherence in patients with COPD. Chest. 2005 Nov;128(5):3198-204. doi: 10.1378/chest.128.5.3198. PMID 16304262
- [Result] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Result] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Result] Oppenheimer BW, Goldring RM, Herberg ME, Hofer IS, Reyfman PA, Liautaud S, Rom WN, Reibman J, Berger KI. Distal airway function in symptomatic subjects with normal spirometry following World Trade Center dust exposure. Chest. 2007 Oct;132(4):1275-82. doi: 10.1378/chest.07-0913. Epub 2007 Sep 21. PMID 17890470
- [Result] Kon SS, Canavan JL, Jones SE, Nolan CM, Clark AL, Dickson MJ, Haselden BM, Polkey MI, Man WD. Minimum clinically important difference for the COPD Assessment Test: a prospective analysis. Lancet Respir Med. 2014 Mar;2(3):195-203. doi: 10.1016/S2213-2600(14)70001-3. Epub 2014 Feb 4. PMID 24621681
- [Result] Han MK, Quibrera PM, Carretta EE, Barr RG, Bleecker ER, Bowler RP, Cooper CB, Comellas A, Couper DJ, Curtis JL, Criner G, Dransfield MT, Hansel NN, Hoffman EA, Kanner RE, Krishnan JA, Martinez CH, Pirozzi CB, O'Neal WK, Rennard S, Tashkin DP, Wedzicha JA, Woodruff P, Paine R 3rd, Martinez FJ; SPIROMICS investigators. Frequency of exacerbations in patients with chronic obstructive pulmonary disease: an analysis of the SPIROMICS cohort. Lancet Respir Med. 2017 Aug;5(8):619-626. doi: 10.1016/S2213-2600(17)30207-2. Epub 2017 Jun 28. PMID 28668356
- [Result] Hogg JC, Chu FS, Tan WC, Sin DD, Patel SA, Pare PD, Martinez FJ, Rogers RM, Make BJ, Criner GJ, Cherniack RM, Sharafkhaneh A, Luketich JD, Coxson HO, Elliott WM, Sciurba FC. Survival after lung volume reduction in chronic obstructive pulmonary disease: insights from small airway pathology. Am J Respir Crit Care Med. 2007 Sep 1;176(5):454-9. doi: 10.1164/rccm.200612-1772OC. Epub 2007 Jun 7. PMID 17556723
- [Result] Basile M, Baiamonte P, Mazzuca E, Principe S, Pennavaria F, Benfante A, Scichilone N. Sleep Disturbances in COPD are Associated with Heterogeneity of Airway Obstruction. COPD. 2018 Jun-Aug;15(4):350-354. doi: 10.1080/15412555.2018.1504015. Epub 2018 Sep 6. PMID 30188194
- [Result] De Backer W, Devolder A, Poli G, Acerbi D, Monno R, Herpich C, Sommerer K, Meyer T, Mariotti F. Lung deposition of BDP/formoterol HFA pMDI in healthy volunteers, asthmatic, and COPD patients. J Aerosol Med Pulm Drug Deliv. 2010 Jun;23(3):137-48. doi: 10.1089/jamp.2009.0772. PMID 20109122
- [Result] de Boer AH, Gjaltema D, Hagedoorn P, Frijlink HW. Can 'extrafine' dry powder aerosols improve lung deposition? Eur J Pharm Biopharm. 2015 Oct;96:143-51. doi: 10.1016/j.ejpb.2015.07.016. Epub 2015 Jul 26. PMID 26220014
- [Result] Virchow JC, Poli G, Herpich C, Kietzig C, Ehlich H, Braeutigam D, Sommerer K, Haussermann S, Mariotti F. Lung Deposition of the Dry Powder Fixed Combination Beclometasone Dipropionate Plus Formoterol Fumarate Using NEXThaler(R) Device in Healthy Subjects, Asthmatic Patients, and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2018 Oct;31(5):269-280. doi: 10.1089/jamp.2016.1359. Epub 2018 Jul 10. PMID 29989511
- [Result] Voshaar T, Spinola M, Linnane P, Campanini A, Lock D, Lafratta A, Scuri M, Ronca B, Melani AS. Comparing usability of NEXThaler((R)) with other inhaled corticosteroid/long-acting beta2-agonist fixed combination dry powder inhalers in asthma patients. J Aerosol Med Pulm Drug Deliv. 2014 Oct;27(5):363-70. doi: 10.1089/jamp.2013.1086. Epub 2013 Dec 3. PMID 24299501
- [Derived] Pisi R, Aiello M, Piraino A, Paleari D, Frizzelli A, Bertorelli G, Chetta A. Beclomethasone/Formoterol in Extra-Fine Formulation Improves Small Airway Dysfunction in COPD Patients. Pulm Ther. 2021 Jun;7(1):133-143. doi: 10.1007/s41030-021-00144-x. Epub 2021 Feb 4. PMID 33538996
- See also: Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2018 — http://goldcopd.org.
- See also: CAT Development Steering Group: COPD Assessment Test - Healthcare Professional User Guide. Issue 4: November 2018. — http://www.catestonline.org